CLINICAL TRIAL: NCT06330233
Title: Construction of Key Technology and Study of the Effect Mechanism of Moxibustion in the Treatment of Diabetic Peripheral Neuropathy Based on Optimal Selection of Acupoints and Moxibustion Volume
Brief Title: Different Amounts of Moxibustion in the Treatment of DPN: A Clinical RCT Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Zhejiang Greentown Cardiovascular Hospital (Other)
Responsible Party: Principal Investigator, Yongliang Jiang, Professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YJiang
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Peripheral Neuropathy; Pain; Moxibustion; Randomized Controlled Trial
Keywords: Diabetic Peripheral Neuropathy; Pain; Moxibustion
MeSH Terms: conditions — Pain | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug treatment group (Sham Comparator): mecobalamin tablets (0.5 mg/dose, 3 times/day) and epalrestat (0.5g/, 3 times/day, before meal) were administered orally for four weeks in conjunction with the patient's daily treatment (basal medication treatment for patients with combined hypertension and hyperlipidemia).
  Interventions: Other: Moxibustion
- Moxibustion 15 minutes group (Experimental): The selected acupoints of moxibustion are Zusanli(ST 36), Sanyinjiao(SP 6), Quchi(LI 11) and Kunlun(BL 60), moxa cones were pasted on the acupoints and moxibustion was applied by ignition, each time for 15 minutes at each acupoint, once every three days, twice a week, four consecutive weeks of treatment.
  Interventions: Other: Moxibustion
- Moxibustion 30 minutes group (Experimental): The selected acupoints of moxibustion are Zusanli(ST 36), Sanyinjiao(SP 6), Quchi(LI 11) and Kunlun(BL 60), moxa cones were pasted on the acupoints and moxibustion was applied by ignition, each time for 30 minutes at each acupoint, once every three days, twice a week, four consecutive weeks of treatment.
  Interventions: Other: Moxibustion

INTERVENTIONS:
Other: Moxibustion — The recruited patients all received diabetes mellitus education. Patients with combined hypertension and hyperlipidemia received daily treatment to lower their blood pressure and blood lipids. The medication was based on their current self-medication, to keep their conditions under normal control. The drug treatment group received mecobalamin tablets and epalrestat orally for four weeks along with their daily treatment. Moxibustion 15-minute group: The selected acupoints of moxibustion are Zusanli(ST 36), Sanyinjiao(SP 6), Quchi(LI 11), and Kunlun(BL 60), moxa cones were pasted on the acupoints and moxibustion was applied by ignition, each time for 15 minutes at each acupoint, once every three days, twice a week, four consecutive weeks of treatment. The moxibustion 30-minute group except for the operating time will use the same intervention as above.

SUMMARY:
This study aims to provide moxibustion treatment for diabetic peripheral neuropathy (DPN) and a reference for clinical treatment of DPN moxibustion. Patients will be randomly assigned to 3 clinical centers, 30 in each center, and then equally divided into 3 groups, including a drug treatment group, a 15-minute moxibustion group, and a 30-minute moxibustion group. Patients in the drug treatment group were given mecobalamin tablets and epalrestat at the same time of daily treatment (hypertension and hyperlipidemia combined with basic drug treatment) for 4 weeks. The frequency of moxibustion was 15/30 minutes per acupoint twice a week for 4 weeks. The results were evaluated during the baseline period (the day before the grouping), the treatment period (the end of the 8th treatment), and the follow-up period (a month after the end of treatment). The results of this part are expected to confirm the therapeutic effect of moxibustion on diabetic peripheral neuropathy. The results of this part will be expected to confirm the optimal amount of moxibustion in the treatment of diabetic peripheral neuralgia and provide a reference for the standardization of clinical treatment of moxibustion.

ELIGIBILITY:
Inclusion Criteria:

1. History of diabetes mellitus;
2. Persistent pain and/or abnormal sensation in the extremities (at least in both lower limbs), decreased bilateral or unilateral ankle reflexes, decreased vibratory sensation (weaker in the medial ankle than in the medial tibial condyle), and decreased nerve conduction velocity on the affected side, and TCSS score >5;
3. 18 years ≤ age ≤ 80 years;
4. Gender is not limited;
5. Those who have the ability of independent daily life and can cooperate to complete all the examinations;
6. Those who are conscious without serious mental diseases and cognitive disorders, and those who do not have serious cardiac, cerebral, hepatic, renal and other internal diseases;
7. Voluntary participation and signing of informed consent.

Exclusion Criteria:

1. Those with peripheral neuropathy, ulcers and gangrene of the limbs caused by various other reasons (e.g. hypothyroidism, alcohol, drugs, heredity, etc.), or those with a history of skin ulcers or lesions that do not heal easily;
2. Women who are in preparation for pregnancy, during pregnancy or breastfeeding;
3. Those with acute complications such as combined diabetic ketoacidosis, lactic acidosis, severe infections, etc.;
4. Those who suffer from serious liver or kidney damage or serious cardiovascular and cerebrovascular diseases (angina pectoris, myocardial infarction, multiple cerebral infarctions, cerebral haemorrhage, etc.);
5. Those who have scars or pigmentation on the skin of the testing site, which will affect the accuracy of the test;
6. Those who are participating in other acupuncture or drug clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total clinical effectiveness | After treatment phase (the 4th week) and the follow-up period (the 5th-8th week)
  Overall clinical effectiveness was assessed at 2 time points: after 4 weeks of treatment and during the follow-up period (the 6th week). It was classified into the following 3 grades according to the Guidelines for Clinical Study of New Chinese Medicines:
  1. Cure: clinical symptoms such as limb numbness, coldness and chilling pain, sensory abnormalities, muscle weakness and muscle atrophy disappear, tendon reflexes return to normal, and the total score of TCSS is ≤ 5 points;
  2. Effective: numbness of the limbs, cold and chilling pain, sensory abnormalities, muscle weakness myasthenia and other clinical symptoms significantly improved, tendon reflexes returned to normal, TCSS score level 2 or 1 level lower;
  3. Ineffective: clinical symptoms did not improve or worsen, tendon reflexes were not elicited, and TCSS score grade did not decrease or increase.
  Total effective rate = [(number of cured cases + number of effective cases)/total number of cases] × 100%.

SECONDARY OUTCOMES:
Electrophysiological examination of the tibial nerve of the lower limb | Baseline (week 0) and the 4th week
  The latency, amplitude, motor nerve conduction velocity (MNCV) and sensory nerve conduction velocity (SNCV) of the tibial nerve of the lower extremities were measured by electrophysiological examination before and after treatment.
Electrophysiological examination of the peroneal nerve of the lower limb | The week 0 and the 4th week
  The latency, amplitude, motor nerve conduction velocity (MNCV) and sensory nerve conduction velocity (SNCV) of the peroneal nerve of the lower extremities were measured by electrophysiological examination before and after treatment.
Toronto Clinical Scoring System | The week 0, the 4th week and the 5th-8th week
  The TCSS is a valid instrument to reflect the presence and severity of diabetic peripheral sensorimotor polyneuropathy as measured by sural nerve morphology and electrophysiology16. TCSS scores of 6-8 for mild DPN, 9-10 for moderate DPN, and 12-19 for sev
Visual Analogue Scale | The week 0, the 4th week and the 5th-8th week
  The level of pain at the subject's lesion site will be determined using the VAS scale, which classifies pain on a scale of 0-10, with the greater the number the more pronounced the pain, i.e., a score of 0 indicates no pain, 2-4 represents mild pain, 5-7 represents moderate pain, 8-9 represents severe pain, and 10 represents severe pain. Allow the subject to indicate the level of pain by crossing out specific numbers on the scale according to their actual situation.
Traditional Chinese Medicine Syndrome Score Scale | The week 0, the 4th week and the 5th-8th week
  The evaluation of the curative effect of TCM symptoms should refer to the guiding principles of clinical research of new drugs of traditional Chinese medicine and the clinical evidence-based practice guide of traditional Chinese medicine for diabetes.
  The specific records are as follows: 1 the VAS score of limb pain was consistent according to the severity. (2) the three main TCM syndromes of limb numbness, abnormal chill (or fever) and ant feeling were scored as 0, 1, 2 and 3 points respectively according to their severity.
infrared thermography testing | The week 0 and the 4th week
  Infrared thermography testing will be performed once before treatment (baseline) and once after 4 weeks of treatment at 2 time points. The test sites will be bilateral plantar, dorsal, palmar, and dorsal hands. The instrument used is the NECR450 infrared thermal imager produced by NECAVIO Company in Japan.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Kang Y, Hu H, Lin C, Zheng Y, Jiang M, Wei Z, He X, Fang J, Jiang Y. Comparative efficacy of moxibustion as an add-on treatment with different durations for diabetic peripheral neuropathy: study protocol for a randomized controlled trial. Front Neurol. 2025 Aug 29;16:1609674. doi: 10.3389/fneur.2025.1609674. eCollection 2025. PMID 40948634